CLINICAL TRIAL: NCT03856970
Title: A Phase 1, Open-Label, Parallel, Sequential, Multi-part Study to Evaluate the Effect of IW-3718 on the Pharmacokinetics of an Oral Contraceptive, Levothyroxine, Glyburide, and Digoxin in Healthy Adult Volunteers
Brief Title: Study to Evaluate the Effect of IW-3718 on the Pharmacokinetics of Oral Contraceptive, Levothyroxine, Glyburide, and Digoxin in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C3718-103
Record Dates: First submitted 2019-02-26; First posted 2019-02-27 (Actual); Last update posted 2019-07-29 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Ethinyl Estradiol; Norethindrone; Thyroxine; Glyburide; Digoxin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Healthy Volunteers (Experimental): Microgestin® (EE 30 μg and NET 1500 μg) single dose (Day 1). After a 10-14 day washout, Microgestin® single dose (Day 14) PLUS IW-3718 1500 mg twice daily (Days 13 to 19).
  Interventions: Drug: Microgestin®; Drug: IW-3718
- Part 2: Healthy Volunteers (Experimental): Levothyroxine 600 μg single dose (Day 1). After a 35-39 day washout, levothyroxine 600 μg single dose (Day 39) PLUS IW-3718 1500 mg twice daily (Days 38 to 41).
  Interventions: Drug: Levothyroxine; Drug: IW-3718
- Part 3: Healthy Volunteers (Experimental): Phase 1: Glyburide 5 mg single dose (Day 1). After a 7-10 day washout, glyburide 5 mg single dose (Day 11) PLUS IW-3718 1500 mg twice daily (ie, Days 10 to 14).
  Phase 2: Digoxin 0.25 mg single dose (Day 23). After a 10-14 day washout, digoxin 0.25 mg mg single dose (Day 35) PLUS IW-3718 1500 mg twice daily (Days 34 to 42).
  Interventions: Drug: Glyburide; Drug: Digoxin; Drug: IW-3718

INTERVENTIONS:
Drug: Microgestin® — 30 μg/1500 μg tablets for oral administration
  Other Names: ethinyl estradiol 30 μg and norethindrone 1500 μg
  Arms: Part 1: Healthy Volunteers
Drug: Levothyroxine — 600 μg tablets for oral administration
  Arms: Part 2: Healthy Volunteers
Drug: Glyburide — 5 mg tablets for oral administration
  Arms: Part 3: Healthy Volunteers
Drug: Digoxin — 0.25 mg tablets for oral administration
  Arms: Part 3: Healthy Volunteers
Drug: IW-3718 — 500-mg film-coated tablets for oral administration

SUMMARY:
The primary objectives of this study are the following:

* To evaluate the pharmacokinetics (PK) of a monophasic oral contraceptive's active components, ethinyl estradiol (EE) and norethindrone acetate (NET), following a single oral dose alone and in combination with IW-3718 in healthy adult female participants.
* To evaluate the PK of levothyroxine following a single oral dose alone and in combination with IW-3718 in healthy adult participants.
* To evaluate the PK of glyburide following a single oral dose alone and in combination with IW-3718 in healthy adult participants.
* To evaluate the PK of digoxin following a single oral dose alone and in combination with IW-3718 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Is healthy, ambulatory, and 18-50 years of age (inclusive) at screening visit.
* Weighs at least 50 kg and has a body mass index within 18-35 kg/m2 at the screening visit.
* Is not pregnant or breastfeeding at the time of the screening visit and has negative serum pregnancy tests at the screening visit and check-in.
* Other inclusion criteria per protocol.

Exclusion Criteria:

* Has used any prescription drugs, herbal supplements, over-the-counter medication, or dietary supplements (vitamins included) within 4 weeks prior to dosing. If needed, (ie, incidental and limited need), acetaminophen is acceptable.
* Has consumed grapefruit or grapefruit juice within 4 weeks prior to dosing or plans to consume grapefruit or grapefruit juice before 7 days following the last dose.
* Has a significant illness that has not resolved within 2 weeks prior to dosing.
* Has a history of immunodeficiency diseases, including a positive human immunodeficiency virus test result.
* Has a positive hepatitis B surface antigen or hepatitis C antibody test result.
* Is a smoker or has used nicotine or nicotine-containing products (eg, snuff, nicotine patch, nicotine chewing gum, mock cigarettes, or inhalers) within 6 months before the first dose of study drug.
* Other exclusion criteria per protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2019-03-11 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-07-03 (Actual)

PRIMARY OUTCOMES:
PK of EE and NET: Area Under the Plasma Concentration Versus Time Curve (AUC) From Time 0 to the Last Quantifiable Concentration (AUC0-t) | Treatment Period 1 (Days 1-6) and Treatment Period 2 (Days 14-19): predose, up to 120 hours postdose
PK of EE and NET: AUC From Time 0 Extrapolated to Infinity (AUC0-inf) | Treatment Period 1 (Days 1-6) and Treatment Period 2 (Days 14-19): predose, up to 120 hours postdose
PK of EE and NET: Maximum Observed Plasma Concentration (Cmax) | Treatment Period 1 (Days 1-6) and Treatment Period 2 (Days 14-19): predose, up to 120 hours postdose
PK of EE and NET: Time to Maximum Observed Plasma Concentration (Tmax) | Treatment Period 1 (Days 1-6) and Treatment Period 2 (Days 14-19): predose, up to 120 hours postdose
PK of EE and NET: Terminal Phase Half-Life (t1/2) | Treatment Period 1 (Days 1-6) and Treatment Period 2 (Days 14-19): predose, up to 120 hours postdose
PK of Levothyroxine: AUC0-t | Treatment Period 1 (Days 1-3) and Treatment Period 2 (Days 39-41): predose, up to 48 hours postdose
PK of Levothyroxine: AUC0-inf | Treatment Period 1 (Days 1-3) and Treatment Period 2 (Days 39-41): predose, up to 48 hours postdose
PK of Levothyroxine: Cmax | Treatment Period 1 (Days 1-3) and Treatment Period 2 (Days 39-41): predose, up to 48 hours postdose
PK of Levothyroxine: Tmax | Treatment Period 1 (Days 1-3) and Treatment Period 2 (Days 39-41): predose, up to 48 hours postdose
PK of Levothyroxine: t1/2 | Treatment Period 1 (Days 1-3) and Treatment Period 2 (Days 39-41): predose, up to 48 hours postdose
PK of Glyburide: AUC0-t | Treatment Period 1 (Days 1-4) and Treatment Period 2 (Days 11-14): predose, up to 72 hours postdose
PK of Glyburide: AUC0-inf | Treatment Period 1 (Days 1-4) and Treatment Period 2 (Days 11-14): predose, up to 72 hours postdose
PK of Glyburide: Cmax | Treatment Period 1 (Days 1-4) and Treatment Period 2 (Days 11-14): predose, up to 72 hours postdose
PK of Glyburide: Tmax | Treatment Period 1 (Days 1-4) and Treatment Period 2 (Days 11-14): predose, up to 72 hours postdose
PK of Glyburide: t1/2 | Treatment Period 1 (Days 1-4) and Treatment Period 2 (Days 11-14): predose, up to 72 hours postdose
PK of Digoxin: AUC0-t | Treatment Period 1 (Days 23-30) and Treatment Period 2 (Days 35-42): predose, up to 168 hours postdose
PK of Digoxin: AUC0-inf | Treatment Period 1 (Days 23-30) and Treatment Period 2 (Days 35-42): predose, up to 168 hours postdose
PK of Digoxin: Cmax | Treatment Period 1 (Days 23-30) and Treatment Period 2 (Days 35-42): predose, up to 168 hours postdose
PK of Digoxin: Tmax | Treatment Period 1 (Days 23-30) and Treatment Period 2 (Days 35-42): predose, up to 168 hours postdose
PK of Digoxin: t1/2 | Treatment Period 1 (Days 23-30) and Treatment Period 2 (Days 35-42): predose, up to 168 hours postdose

SECONDARY OUTCOMES:
Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs), and Discontinuations due to TEAEs | Part 1: up to Day 27 (±1 day); Part 2: up to Day 49 (±1 day); Part 3: Day 50 (±1 day)
Number of Participants With ≥1 Clinically Significant Changes in Clinical Laboratory Test Results | Part 1: up to Day 19; Part 2: up to Day 41; Part 3: up to Day 42
Number of Participants With ≥1 Clinically Significant Changes in Vital Sign Measurements | Part 1: up to Day 19; Part 2: up to Day 41; Part 3: up to Day 42
Number of Participants With ≥1 Clinically Significant Changes in 12-lead Electrocardiogram (ECG) Results | Part 1: up to Day 19; Part 2: up to Day 41; Part 3: up to Day 42
Number of Participants With ≥1 Clinically Significant Changes in Physical Examination Findings | Part 1: up to Day 19; Part 2: up to Day 41; Part 3: up to Day 42

CONTACTS AND LOCATIONS:
Overall Officials: Zurab Machaidze, MD, Study Director — Ironwood Pharmaceuticals, Inc.
Locations (1):
- PPD, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided